CLINICAL TRIAL: NCT06623084
Title: Integrated Phenotyping of the Gut-plAtelet-Liver AXIS in the Progression of Chronic Liver Disease (iGAL-AXIS)
Status: Not yet recruiting | Type: Observational
Sponsor: Stefania Basili (Other)
Collaborators: University of Rome Tor Vergata (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor-Investigator, Stefania Basili, Head of Internal medicine Stefania Basili, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: 6804
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); NASH - Nonalcoholic Steatohepatitis; Cirrhosis; Control Condition
Keywords: Platelets; Liver; Metabolomics; Microbiota
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The investigators plan to recruit n=33 subjects with NAFLD, n=33 subjects with histologically proven NASH and n=33 subjects with metabolic non-viral cirrhosis and n=33 sex- and age-matched metabolically healthy volunteers (without NAFLD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- NAFL GROUP: The investigators plan to recruit n=33 subjects with NAFLD
  Interventions: Other: Platelets characterization
- NASH GROUP: The investigators plan to recruit n=33 subjects with histologically proven NASH
  Interventions: Other: Platelets characterization
- Cirrhotic patients: The investigators plan to recruit n=33 subjects with metabolic non-viral cirrhosis
  Interventions: Other: Platelets characterization
- Controls group: The investigators plan to recruit n=33 sex- and age-matched metabolically healthy volunteers (without NAFLD)
  Interventions: Other: Platelets characterization

INTERVENTIONS:
Other: Platelets characterization — To identify platelet features that correlate with liver disease progression and to study the mechanistic relationship between gut dysbiosis, metabolome composition, inflammation, and platelet activation in chronic liver disease.

SUMMARY:
Objective of the study Our working hypothesis is that platelets activated by gut-derived metabolites dock in the liver of NAFLD patients and amplify the inflammatory state by releasing pro-inflammatory cytokines/chemokines, which in turn recruit and activate leukocytes in the liver sinusoids. Combined stimuli from leukocytes and platelets would then lead to metabolic reprogramming of hepatocytes, progression to NASH and eventually cirrhosis.

To test this hypothesis, the investigators propose 2 objectives. Primary objective: To identify platelet features that correlate with liver disease progression.

Secondary objective: To study the mechanistic relationship between gut dysbiosis, metabolome composition, inflammation, and platelet activation in chronic liver disease.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the main cause of chronic liver diseases and is now considered a global health problem. NAFLD is a spectrum of diseases ranging from simple hepatic steatosis (NAFL) to non-alcoholic Steatohepatitis (NASH). Over time, NAFLD may progress to cirrhosis and ultimately to hepatocellular carcinoma (HCC). The gold-standard for diagnosis is liver biopsy that allows to discriminate different types of steatosis, characterized by the accumulation of lipid droplets of different sizes in hepatocytes, with the largest droplets associated with the development of fibrosis and the severity of the disease. Future studies are needed to identify non- invasive diagnostic approaches alternative to liver biopsy. NAFLD is not considered a "hepato-centric" condition anymore. Bi-directional metabolic and immune lanes of communication with other organs, such as the gut, have been decoded. Gut dysbiosis, increased gut permeability and bacterial translocation within portal circulation have been reported in NAFLD, suggesting that the gut-liver axis represents a source of systemic and hepatic inflammation.

Many studies suggest that platelets may be the link between gut and liver dysfunction. Beyond their role in hemostasis platelets can sense PAMPs and DAMPs and actively participate in the inflammatory response and in tissue remodeling, by releasing bioactive molecules and by interacting with leukocytes. Gut-derived metabolites and bacterial endotoxins promote platelet hyper-reactivity and recent studies point to an important role of platelets in regulating chronic liver inflammation. Platelet-derived cytokines, such as TGF-β, PDGF-β and CXCL4 promote hepatic fibrosis, and platelet count has been used as a surrogate marker of liver fibrosis FIB-4 index). Platelet number and platelet aggregates are increased in liver sinusoids of NASH patients and colocalise with neutrophil extracellular traps (NETs). In mice it was shown that platelet colonization of the liver is a critical step for the recruitment of CD8+ T cells and NKT cells, which drive NASH progression through the release of cytokines and the metabolic reprogramming of hepatocytes. In humans, inhibition of platelets with a combination of aspirin and clopidogrel has been shown to reduce the development of NASH and subsequent progression to cirrhosis and HCC. Mechanistic insights suggest that the role of platelets in NAFLD progression is mediated through the interaction with immune cells.

ELIGIBILITY:
Inclusion Criteria:

* age>18;
* NAFLD patients according to EASL Guidelines 2016.

Exclusion Criteria:

* decompensated cirrhosis, other causes of chronic liver disease (infectious and immune-mediated); malabsorption syndromes (i.e., celiac disease, food allergy, small bowel bacterial overgrowth);
* inflammatory bowel disease; previous GI surgery;
* immunodeficiencies; neurological handicaps;
* use of NSAIDs, antibiotics, probiotics, or anti-secretory drugs within the 2 months preceding enrollment;
* abnormality of hemostasis and thrombosis; malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 132 individuals (n=33 subjects with NAFLD, n=33 subjects with histologically proven NASH and n=33 subjects with metabolic non-viral cirrhosis and n=33 healthy volunteers (without NAFLD) will be enrolled at the Policlinico Umberto I-Sapienza University of Rome, defined according to the EASL Guidelines 2016.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-03-12 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Inflammatory profiling | 1 year
  To compare the systemic inflammatory state of patients at different stages of liver disease, serum samples will be used to quantify the concentration of 13 inflammatory cytokines (pg/ml), including IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, and IL-33, by multiplex bead-based flow cytometric assay. Moreover, serum samples will be analysed by standard ELISA for the presence of HMGB1 and calprotectin (MRP8/14), inflammatory biomarkers that are associated with liver disease progression, and for the presence of DNA-myeloperoxidase complexes that are specific markers of neutrophil extracellular traps (NETs).

IPD SHARING:
Plan to Share IPD: No